CLINICAL TRIAL: NCT06301971
Title: A Phase 1, Open-Label Trial to Assess the Mass Balance, Pharmacokinetics, Metabolism, and Excretion of Emraclidine in Healthy Adult Male Participants
Brief Title: A Study to Assess Mass Balance, Pharmacokinetics, Metabolism, and Excretion of Emraclidine in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-HV-1011
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emraclidine 30 mg (Experimental): Participants will receive a single oral dose of 30 milligrams (mg) (approximately 75 microcurie [μCi]) [14C]-emraclidine on Day 1.
  Interventions: Drug: Emraclidine

INTERVENTIONS:
Drug: Emraclidine — Oral solution/suspension
  Other Names: CVL-231

SUMMARY:
The primary purpose of this study is to determine the mass balance, routes, and rates of elimination of total radioactivity and characterize the pharmacokinetics (PK) of emraclidine, metabolite CV-0000364, and total radioactivity in plasma and whole blood following a single oral dose of [14C]-emraclidine in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) of 18.5 to 35.0 kilograms per square meters (kg/m^2), inclusive, and a total body weight ≥50 kg [110 Pounds (lbs)].
2. A male participant who is sexually active with a pregnant or a nonpregnant woman of childbearing potential must agree to use a condom during the trial and for 90 days after the dose of investigational medicinal product (IMP). In addition, male participants should not donate sperm for a minimum of 90 days following the dose of IMP.
3. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.
4. Capable of consuming the standard diet.
5. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

   * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
   * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior)

   "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
   * Suicidal Ideation Item 1 (Wish to be Dead)
   * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary.
3. Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
4. Use of any prescription and over-the-counter medications from 28 days prior to first dose of IMP or likely to require concomitant therapy. Vaccinations or boosters within 28 days of planned dosing or while on trial.
5. Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B total core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
6. Positive drug screen (including cotinine and tetrahydrocannabinol [THC]) or a positive test for alcohol.
7. Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement, if deemed necessary:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2× upper limit of normal (ULN).
   * Total bilirubin ≥1.5×ULN. If Gilbert's syndrome is suspected, total bilirubin ≥1.5×ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.
8. Known allergy or hypersensitivity to the IMP, closely related compounds, or any of their specified ingredients.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — U.S. Food and Drug Administration (FDA) recommends that radiation exposure to participants should be kept as low as is reasonably achievable; and since there is no available data to suggest metabolism of the emraclidine is different in women versus men. Hence, female participants are excluded from this study.
Enrollment: 8 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Curve (AUC) from Zero to Infinity (AUCinf) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
AUC from Time 0 to last Quantifiable Concentration (AUClast) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Maximum Plasma Concentration (Cmax) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Time to Last Measurable Concentration (Tlast) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Time to Maximum Observed Concentration (Tmax) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Apparent Terminal Elimination Half-life (t½) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Terminal Rate Constant (λz) of Emraclidine, its Metabolite CV-0000364 and Total Radioactivity in Plasma and Whole Blood | Pre-dose and at multiple time points post-dose up to Day 15
Total Plasma Clearance After Oral Administration (CL/F) of Emraclidine | Pre-dose and at multiple time points post-dose up to Day 15
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Emraclidine | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Plasma AUCinf for Emraclidine to Plasma AUCinf for Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Plasma AUCinf for Metabolite CV-0000364 to Plasma AUCinf for Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Plasma AUCinf for Metabolite CV-0000364 to Plasma AUCinf for Emraclidine | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Whole Blood AUCinf for Total Radioactivity to Plasma AUCinf for Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Amount Excreted in Urine (Aeu) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Cumulative Aeu of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Percentage Excreted in Urine (feu) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Cumulative feu of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Amount Excreted in Feces (Aef) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Cumulative Aef of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Percentage Excreted in Feces (fef) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Cumulative fef of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Percentage Dose (%Dose) of Total Radioactivity Excreted in Urine Plus Feces Combined | Pre-dose and at multiple time points post-dose up to Day 15
Cumulative Percentage Dose of Total Radioactivity Excreted in Urine Plus Feces Combined | Pre-dose and at multiple time points post-dose up to Day 15

SECONDARY OUTCOMES:
Metabolite Profile of Emraclidine in Plasma, Urine and Feces | Pre-dose and at multiple time points post-dose up to Day 15
Structural Identification of Emraclidine Metabolites Found in Plasma, Urine and Feces | Pre-dose and at multiple time points post-dose up to Day 15
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 16
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 15
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 15
Number of Participants with Clinically Significant Changes in Laboratory Assessments | Up to Day 15
Number of Participants with Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 15
Change from Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Day 15
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No